CLINICAL TRIAL: NCT02351401
Title: Improvement in Patient Awareness and Ability to Assess Disease in Rheumatoid Arthritis: Rheumatoid Arthritis Through Education and US Study (RAEUS)
Brief Title: Rheumatoid Arthritis Through Education and US Study (RAEUS)
Acronym: RAEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Medicine, Dr Peter Cheung, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011/01611
Record Dates: First submitted 2015-01-12; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education with ultrasonography (Experimental): Intervention includes education of self-assessment of synovitis using ultrasonography as a feedback training tool
  Interventions: Behavioral: Education using ultrasonography as feedback tool
- Standard Care (No Intervention): Normal standard care where patients are not taught how to self-assess for synovitis, without ultrasonography a training tool

INTERVENTIONS:
Behavioral: Education using ultrasonography as feedback tool — Education using ultrasonography as feedback tool
  Arms: Education with ultrasonography

SUMMARY:
Patients can potentially monitor disease activity of rheumatoid arthritis (RA) through self-assessed swollen joints (clinical synovitis)joint counts but reliability of joint swelling is poor. The objective is to evaluate the use of education by ultrasound feedback on the ability of patients to assess for clinical synovitis swollen joints in RA.

DETAILED DESCRIPTION:
Design: 6-month single centre randomized controlled trial. Patients: established RA. Intervention: education on self-assessment of joints that included initial brief patient training on tender (TJC) and swollen (SJC) joint counts, followed by US feedback every 3 months versus standard care without education. Patient and physician independently performed 28-joint counts at each visit. Outcome variables: (Primary) Percentage of patients with good agreement with physician derived swollen joints (prevalence-adjusted bias adjusted kappa, PABAK>0.6). Other variables: Agreement in SJC (Bland and Altman 95% limits of agreement), feasibility/patient satisfaction survey and disease activity score (DAS28) at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* RA patients fulfilling ACR1987 criteria
* adults between age 21 and 80 years

Exclusion Criteria:

* pregnant
* no mental health illness
* fit to perform informed consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
prevalence-adjusted bias adjusted kappa, PABAK>0.6 | at 6 months

SECONDARY OUTCOMES:
Bland and Altman 95% limits of agreement | 6 months
  swollen joint count agreement
Level of satisfaction | 6 months
  Likert response, satisfaction survey
disease activity score in 28 joints (DAS28) | 6 months
  composite score that measures disease activity incorporating tender joint count, swollen joint count, erythrocyte sedimentation rate and patient global assessment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cheung, Principal Investigator — National University Hospital, Rheumatology

REFERENCES:
- [Derived] Cheung PP, Lahiri M, Teng GG, Lim AY, Lau TC, Lateef A, Mak A, Gossec L, March L. A randomized controlled trial for improving patient self-assessment of synovitis in rheumatoid arthritis with education by ultrasonography: the RAEUS Study. Rheumatology (Oxford). 2015 Jul;54(7):1161-9. doi: 10.1093/rheumatology/keu447. Epub 2014 Dec 3. PMID 25477057